CLINICAL TRIAL: NCT06837714
Title: Investigation of the Effects of Pilates Exercises on Menopausal Symptoms and Sexual Dysfunction in Postmenopausal Women
Brief Title: Investigation of the Effects of Pilates Exercises on Menopause Symptoms and Sexual Dysfunction in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Batman University (Other)
Responsible Party: Principal Investigator, merve yiğit kocamer, lecturer, Batman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAU-FTR-MYK-01
Record Dates: First submitted 2024-12-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Menopausal Syndrome; Sexual Dysfunctions; Quality of Life and Menopause
Keywords: postmenopause; pilates; menopausal syndrome; sexual dysfunctions; Quality of life

STUDY DESIGN:
Intervention Model Description: 1. Reformer pilates group
  2. Group that includes lifestyle changes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pilates group (Active Comparator): The Pilates intervention group participated in an 8-week Pilates exercise program. The program consisted of sessions held twice a week, each lasting approximately 60 minutes. The Pilates exercises focused on core stability, flexibility, balance, and controlled breathing, and were tailored to accommodate the fitness levels of the participants. Each session was conducted by a certified Pilates instructor who ensured proper technique and safety during the exercises
  Interventions: Other: PİLATES GROUP
- group that includes lifestyle changes (Active Comparator): . The control group did not engage in any structured exercise program during the 8-week period. Instead, they attended a menopause information session where they received education on menopause-related issues, including symptom management, lifestyle modifications, and general health tips for postmenopausal women.
  Interventions: Other: Behavioral: lifestyle changes

INTERVENTIONS:
Other: PİLATES GROUP — A total of 16 sessions were applied for 8 weeks, 2 sessions per week.
  Arms: pilates group
Other: Behavioral: lifestyle changes — presentation including lifestyle changes was prepared and training was provided.
  Arms: group that includes lifestyle changes

SUMMARY:
Menopause represents a major transition in a woman's life as estrogen and progesterone levels decline, and this hormonal shift is associated with a range of symptoms that can significantly impact a woman's quality of life, including vasomotor symptoms such as hot flushes and night sweats, and urogenital symptoms such as vaginal dryness and sexual dysfunction.

DETAILED DESCRIPTION:
This study aimed to investigate the effects of Pilates exercises on menopausal symptoms and sexual dysfunction in postmenopausal women. The research seeks to understand how an 8-week Pilates program, conducted twice a week, influences the quality of life and sexual function during the postmenopausal period. A total of 30 postmenopausal women were included in this study, divided into a Pilates group and a control group. The Pilates group participated in an 8-week Pilates exercise program, while the control group received no exercise intervention but attended menopause information sessions. Data were collected using the Menopause Rating Scale (MRS), the Menopausal-Specific Quality of Life Scale (MENQOL), and the Female Sexual Function Index (FSFI) before and after the intervention. Body Mass Index (BMI) was recorded, but not used in the primary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women who have reached menopause
* Being physically or cognitively competent to exercise
* Those who agreed to participate in the study

Exclusion Criteria:

* Those with serious heart disease, DM, kidney, liver, thyroid disease and cancer patients
* Those receiving hormone therapy
* People using antipsychotic medication
* Those using steroids and derivative drugs
* People using insulin sensitizing drugs Those with musculoskeletal system diseases that would prevent them from exercising Cognitive problems that affect cooperation

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 30 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Menopause Rating Scale (MRS) | 8 week
  This scale was used to assess the severity of menopausal symptoms experienced by the participants. The MRS covers a range of symptoms, including vasomotor, psychological, and urogenital symptoms. Participants rated the severity of each symptom on a Likert scale, with higher scores indicating more severe symptoms. The total score of the scale is calculated with the scores obtained from each item. The lowest score calculated from the scale is "0" while the highest score is "44". The scale covering menopausal symptoms consists of 11 items and 3 sub-dimensions. The sub-dimensions are somatic complaints (items 1, 2, 3 and 11), psychological complaints (items 4, 5, 6 and 7), urogenital complaints (items 8, 9 and 10). An increase in the total score obtained from the scale indicates an increase in the severity of the complaints experienced and, in addition, a negative impact on the quality of life.
Menopausal-Specific Quality of Life Scale (MENQOL) | 8 week
  This scale measures the impact of menopausal symptoms on quality of life across several domains, including physical, psychological, and sexual well-being. The MENQOL provides a comprehensive assessment of how menopausal symptoms affect daily life, with higher scores indicating a greater negative impact.MENQOL is a Likert-type scale containing 32 questions. It consists of four sub-areas: vasomotor, psychosocial, physical and sexual. Each sub-area score in MENQOL is ranked from 1 to 8. A score of one indicates that no problem is experienced regarding that issue, a score of two indicates that the issue exists, is experienced but is not disturbing at all, while scores between 3 and 8 indicate the severity and increasing degrees of the existing problem. The maximum score is 256, and the minimum score is 32.
Female Sexual Function Index (FSFI) | 8 week
  The FSFI was used to evaluate sexual function, focusing on domains such as sexual desire, arousal, lubrication, orgasm, satisfaction, and pain. Participants were asked to rate their experiences in each domain over the past 4 weeks. Higher FSFI scores indicate better sexual function.The highest raw score that can be obtained from the survey is 95, and the lowest is 4. The total score obtained from the survey shows that there is an improvement in all parameters as the scores obtained from the parameters of sexual desire, arousal, lubrication, orgasm, and general satisfaction increase.

CONTACTS AND LOCATIONS:
Overall Officials: YİĞİT KOCAMER MERVE, Principal Investigator — Batman University
Locations (3):
- Turkey (Türkiye) (3):
  - Batman Center, Batman, Gültepe
  - Batman university, Batman
  - Türkiye, Batman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yigit Kocamer M, Atilgan E. Investigating the effects of Pilates exercises on menopausal symptoms and sexual dysfunction in postmenopausal women: A randomized controlled trial. Medicine (Baltimore). 2025 Jun 6;104(23):e42689. doi: 10.1097/MD.0000000000042689. PMID 40489883